CLINICAL TRIAL: NCT01267604
Title: Improving Oocyte Retrieval Using a Combined Therapy of Recombinant Follicle Stimulating Hormone (rFSH) and Inositol and Melatonin
Brief Title: Ovarian Stimulation: Inositol and Melatonin
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Collaborators: University of Modena and Reggio Emilia (Other); Research Center for Reproductive Medicine Villa Mafalda (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rFSH-INOPLUS
Record Dates: First submitted 2010-12-23; First posted 2010-12-28 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Inositol; Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recombinant FSH (Active Comparator): 225IU rFSH
  Interventions: Drug: Recombinant FSH (rFSH)
- Recombinant FSH Inositol Melatonin (Experimental): 225IU rFSH, 4g Inositol and 3mg Melatonin
  Interventions: Dietary Supplement: rFSH + Inositol + Melatonin

INTERVENTIONS:
Drug: Recombinant FSH (rFSH) — 225IU
  Arms: Recombinant FSH
Dietary Supplement: rFSH + Inositol + Melatonin — 225IU rFSH, 4g Inositol, 3mg Melatonin
  Arms: Recombinant FSH Inositol Melatonin

SUMMARY:
An efficient protocol of ovarian stimulation is a key part of assisted reproductive technology. In order to obtain the highest oocyte retrieval with no adverse effects, numerous studies have evaluated the efficiency of the clinical approaches currently available.

Recent studies have shown that two natural compounds, such as inositol and melatonin, play an important role in oocyte maturation and quality. Therefore, the present study aims at investigating whether inositol and melatonin are able to improve the number of oocytes obtained after ovarian stimulation with Recombinant Follicle Stimulating Hormone (rFSH).

To this purpose, a randomized double-blind trial will be established where 150 healthy women in reproductive age undergoing to assistant reproductive technology (ART) because of male infertility will be divided in two groups. Group A will be treated with 225IU rFSH alone, group B will be treated with 225IU rFSH, 4g inositol and 3mg melatonin.

As primary outcome of the study, oocyte quality, total number of oocytes retrieved, clinical pregnancy rate and live birth rate will be evaluated in group A vs. group B.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18-39 years
* BMI 18-30 kg/m2,
* Fewer than 3 prior oocyte retrievals,
* No fertility Problems

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Total oocyte number | 2 weeks after pharmacological treatment
Number of clinical pregnancies | 6 weeks after embryo transfer
Live birth rate | 10 months after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Unfer, MD, Study Director — AGUNCO Obstetrics and Gynecology Centre; Gianfranco Carlomagno, PhD, Principal Investigator — AGUNCO Obstetrics and Gynecology Centre; La Sala Giovanni Battista, MD, Principal Investigator — University of Modena and Reggio Emilia; Franco Lisi, MD, Principal Investigator — Research Center for Reproductive Medicine
Locations (2):
- Italy (2):
  - University of Modena and Reggio Emilia, Reggio Emilia
  - Research Center for Reproductive Medicine Villa Mafalda, Roma

REFERENCES:
- [Background] Rizzo P, Raffone E, Benedetto V. Effect of the treatment with myo-inositol plus folic acid plus melatonin in comparison with a treatment with myo-inositol plus folic acid on oocyte quality and pregnancy outcome in IVF cycles. A prospective, clinical trial. Eur Rev Med Pharmacol Sci. 2010 Jun;14(6):555-61. PMID 20712264
- [Background] Papaleo E, Unfer V, Baillargeon JP, Chiu TT. Contribution of myo-inositol to reproduction. Eur J Obstet Gynecol Reprod Biol. 2009 Dec;147(2):120-3. doi: 10.1016/j.ejogrb.2009.09.008. Epub 2009 Oct 2. PMID 19800728
- [Background] Tamura H, Nakamura Y, Korkmaz A, Manchester LC, Tan DX, Sugino N, Reiter RJ. Melatonin and the ovary: physiological and pathophysiological implications. Fertil Steril. 2009 Jul;92(1):328-43. doi: 10.1016/j.fertnstert.2008.05.016. Epub 2008 Sep 18. PMID 18804205